CLINICAL TRIAL: NCT02151110
Title: A Phase 1, Randomized, Blinded, Placebo-controlled, Single-ascending Dose Study to Evaluate the Safety and Tolerability of MEDI4920 in Healthy Adults
Brief Title: Phase 1 Single-ascending Dose Study to Evaluate Safety and Tolerability of MEDI4920 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5100C00001
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Healthy Volunteer
Keywords: Healthy Male; Healthy Female of non child bearing potential

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Placebo (Placebo Comparator): Participants received single IV dose of placebo matching with MEDI4920 infused on Day 1.
  Interventions: Other: Placebo
- MEDI4920 3 mg (Experimental): Participants received single IV dose of MEDI4920 3 milligram (mg) infused on Day 1.
  Interventions: Biological: MEDI4920 3 mg
- MEDI4920 10 mg (Experimental): Participants received single IV dose of MEDI4920 10 mg infused on Day 1.
  Interventions: Biological: MEDI4920 10 mg
- MEDI4920 30 mg (Experimental): Participants received single IV dose of MEDI4920 30 mg infused on Day 1.
  Interventions: Biological: MEDI4920 30 mg
- MEDI4920 100 mg (Experimental): Participants received single IV dose of MEDI4920 100 mg infused on Day 1.
  Interventions: Biological: MEDI4920 100 mg
- MEDI4920 300 mg (Experimental): Participants received single IV dose of MEDI4920 300 mg infused on Day 1.
  Interventions: Biological: MEDI4920 300 mg
- MEDI4920 1000 mg (Experimental): Participants received single IV dose of MEDI4920 1000 mg infused on Day 1.
  Interventions: Biological: MEDI4920 1000 mg
- MEDI4920 3000 mg (Experimental): Participants received single IV dose of MEDI4920 3000 mg infused on Day 1.
  Interventions: Biological: MEDI4920 3000 mg

INTERVENTIONS:
Biological: MEDI4920 3 mg — Participants received single IV dose of MEDI4920 3 milligram (mg) infused on Day 1.
  Arms: MEDI4920 3 mg
Biological: MEDI4920 10 mg — Participants received single IV dose of MEDI4920 10 mg infused on Day 1.
  Arms: MEDI4920 10 mg
Biological: MEDI4920 30 mg — Participants received single IV dose of MEDI4920 30 mg infused on Day 1.
  Arms: MEDI4920 30 mg
Biological: MEDI4920 100 mg — Participants received single IV dose of MEDI4920 100 mg infused on Day 1.
  Arms: MEDI4920 100 mg
Biological: MEDI4920 300 mg — Participants received single IV dose of MEDI4920 300 mg infused on Day 1.
  Arms: MEDI4920 300 mg
Biological: MEDI4920 1000 mg — Participants received single IV dose of MEDI4920 1000 mg infused on Day 1.
  Arms: MEDI4920 1000 mg
Biological: MEDI4920 3000 mg — Participants received single IV dose of MEDI4920 3000 mg infused on Day 1.
  Arms: MEDI4920 3000 mg
Other: Placebo — Participants received single IV dose of placebo matching with MEDI4920 infused on Day 1.
  Arms: Placebo

SUMMARY:
Phase 1 single IV dose study to evaluate safety and tolerability of MEDI4920

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible study physician based on medical evaluation
* Body weight 40 to 100 kg
* Body mass index 19.0 to 30.0 kg/m2

Exclusion Criteria:

* History of allergy or sensitivity to Shellfish or protein based antigens
* previous immunization with KLH
* previous splenectomy
* History of diagnosed or suspected thromboembolic event or coagulation disorder

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2016-05-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Leeds, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult male and female participants were recruited in a blinded manner. The study was conducted at one site in the United Kingdom.
Pre-assignment Details: A total of 259 participants were screened of which 200 participants were considered screen failures and the remaining 59 participants were randomized. Out of which, 56 participants were treated
Period: Overall Study
Arm/Group | Placebo | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Started | 12 | 2 | 2 | 8 | 8 | 8 | 8 | 8
Completed | 12 | 2 | 2 | 8 | 8 | 8 | 8 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any study drug. Two participants were erroneously randomized to MEDI4920 10 mg group due to the IXRS system not being opened for start of MEDI4920 30 mg group. However, these participants received the 30 mg dose.
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | Placebo | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg | TOTAL
Number analyzed (Participants) | 12 | 2 | 2 | 8 | 8 | 8 | 8 | 8 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.3 (8.9) | 27.5 (4.9) | 26.0 (1.4) | 27.8 (12.3) | 28.1 (10.1) | 38.4 (9.3) | 33.3 (9.2) | 32.0 (9.8) | 31.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 12 | 2 | 2 | 8 | 8 | 8 | 8 | 8 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening situation (immediate risk of dying); persistent or significant disability or incapacity; congenital anomaly or birth defect in the offspring of a participant who received the study drug. A TEAE is defined as the event with onset after the start of infusion (Day 1) to Day 113 or early discontinuation visit inclusive. The AEs were summarized using Medical Dictionary for Regulatory Activities version 19.0.
Time Frame: The start of study drug administration (Day 1) to the follow-up period (Day 113) or early discontinuation visit
Population: As-treated Population: All participants who received any study drug were included in this population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Number analyzed (Participants) | 12 | 2 | 2 | 8 | 8 | 8 | 8 | 8
Participants
  TEAEs | 10 | 1 | 1 | 5 | 8 | 3 | 5 | 7
  TESAEs | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MEDI4920
Description: The maximum observed plasma concentration (Cmax) was estimated based on the plasma concentrations of MEDI4920. Standard deviation was calculated only if number of participants were more than or equal to 3.
Time Frame: Pre-infusion, at the middle of the infusion, post-infusion (5 minutes, and 2, 6, and 12 hours) on Day 1; Days 2, 3, 5, 8, 15, 22, 29, 43, 57, 85, and 113 or early discontinuation visit, whichever occurred first
Population: As-treated Population
Measure: Mean (Standard Deviation); unit: microgram per milliliter (µg/mL)
Arm/Group | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Number analyzed (Participants) | 2 | 2 | 8 | 8 | 8 | 8 | 8
microgram per milliliter (µg/mL) | 1.00 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 4.46 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 7.97 (0.873) | 23.6 (2.76) | 85.6 (17.6) | 289 (58.1) | 960 (126)

3. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-last) of MEDI4920
Description: The area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last) was estimated based on the plasma concentrations of MEDI4920. Standard deviation was calculated only if number of participants were more than or equal to 3.
Time Frame: as for outcome 2
Population: As-treated Population
Measure: Mean (Standard Deviation); unit: microgram*day per milliliter (µg*d/mL)
Arm/Group | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Number analyzed (Participants) | 2 | 2 | 8 | 8 | 8 | 8 | 8
microgram*day per milliliter (µg*d/mL) | 3.64 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 19.3 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 53.4 (10.9) | 151 (20.2) | 581 (38.3) | 2090 (394) | 6640 (553)

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of MEDI4920
Description: The area under the plasma concentration-time curve from time zero to infinity (AUC 0-inf) was estimated based on the plasma concentrations of MEDI4920. Standard deviation was calculated only if number of participants were more than or equal to 3.
Time Frame: as for outcome 2
Population: As-treated Population
Measure: Mean (Standard Deviation); unit: microgram*day per milliliter (µg*d/mL)
Arm/Group | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Number analyzed (Participants) | 2 | 2 | 8 | 8 | 8 | 8 | 8
microgram*day per milliliter (µg*d/mL) | 4.60 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 20.5 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 54.8 (11.0) | 152 (20.2) | 583 (37.8) | 2090 (394) | 6640 (547)

5. Secondary Outcome: Dose-normalized AUC0-inf (AUC0-infinity/D) of MEDI4920
Description: The AUC (0-infinity)/D is the area under concentration-time curve extrapolated to infinity postdose normalized by MEDI4920 dose. The AUC (0-infinity)/D was estimated based on the plasma concentrations of MEDI4920. Standard deviation was calculated only if number of participants were more than or equal to 3.
Time Frame: as for outcome 2
Population: As-treated Population
Measure: Mean (Standard Deviation); unit: µg*d/mL/mg
Arm/Group | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Number analyzed (Participants) | 2 | 2 | 8 | 8 | 8 | 8 | 8
µg*d/mL/mg | 1.53 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 2.05 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 1.83 (0.366) | 1.52 (0.202) | 1.94 (0.126) | 2.09 (0.394) | 2.21 (0.182)

6. Secondary Outcome: Terminal Elimination Half Life (t1/2) of MEDI4920
Description: The terminal elimination half-life (t1/2) was estimated based on the plasma concentrations of MEDI4920. Standard deviation was calculated only if number of participants were more than or equal to 3.
Time Frame: as for outcome 2
Population: As-treated Population
Measure: Mean (Standard Deviation); unit: Day(s)
Arm/Group | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Number analyzed (Participants) | 2 | 2 | 8 | 8 | 8 | 8 | 8
Day(s) | 4.41 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 5.35 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 5.31 (2.30) | 5.49 (1.59) | 8.86 (1.60) | 9.68 (1.25) | 10.1 (1.87)

7. Secondary Outcome: Systemic Clearance (CL) of MEDI4920
Description: The systemic clearance (CL) was estimated based on the plasma concentrations of MEDI4920. Standard deviation was calculated only if number of participants were more than or equal to 3.
Time Frame: as for outcome 2
Population: As-treated Population
Measure: Mean (Standard Deviation); unit: milliliter per day (mL/day)
Arm/Group | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Number analyzed (Participants) | 2 | 2 | 8 | 8 | 8 | 8 | 8
milliliter per day (mL/day) | 661 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 487 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 564 (96.8) | 668 (90.4) | 517 (33.5) | 494 (102) | 454 (37.9)

8. Secondary Outcome: Volume of Distribution at Steady-state (Vss) of MEDI4920
Description: The volume of distribution at steady-state (Vss) was estimated based on the plasma concentrations of MEDI4920. Standard deviation was calculated only if number of participants were more than or equal to 3.
Time Frame: as for outcome 2
Population: As-treated Population
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Number analyzed (Participants) | 2 | 2 | 8 | 8 | 8 | 8 | 8
milliliter (mL) | 3980 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 3290 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 4280 (684) | 5560 (806) | 5180 (811) | 5450 (1150) | 4900 (715)

9. Secondary Outcome: Volume of Distribution Based on Terminal Phase (Vz) of MEDI4920
Description: The volume of distribution based on terminal phase (Vz) was estimated based on the plasma concentrations of MEDI4920. Standard deviation was calculated only if number of participants were more than or equal to 3.
Time Frame: as for outcome 2
Population: As-treated Population
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Number analyzed (Participants) | 2 | 2 | 8 | 8 | 8 | 8 | 8
milliliter (mL) | 4130 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 3760 (NA) — Not calculated; Standard deviation was only calculated if N >= 3. | 4080 (1090) | 5230 (1360) | 6590 (1160) | 6880 (1520) | 6600 (1190)

10. Secondary Outcome: Percentage of Participants Positive for Anti-drug Antibodies (ADA)
Description: Plasma samples were collected for assessment of anti-drug antibodies (ADA) against MEDI4920. The incidence of positive serum antibodies to MEDI4920 are presented.
Time Frame: Baseline (pre-infusion on Day 1) and post-baseline Days 15, 29, 57, and 113 or early discontinuation visit, whichever occurred first
Population: As-treated Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Number analyzed (Participants) | 12 | 2 | 2 | 8 | 8 | 8 | 8 | 8
Percentage of participants
  Baseline ADA positive | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post-baseline ADA positive | 8.3 | 50 | 100 | 100 | 87.5 | 37.5 | 37.5 | 12.5

11. Secondary Outcome: T-cell Dependent Antibody Response (TDAR) Measured by Anti-keyhole Limpet Hemocyanin Immunoglobulin G (Anti-KLH IgG) Concentration
Description: The T-cell dependent antibody response (TDAR) assay measures the immune response (ie, antibody production) to an introduced antigen, keyhole limpet hemocyanin (KLH). The KLH is a potent immunostimulating protein with an extensive history of safe and effective use in vaccine development and immunological research. TDAR was evaluated by measuring anti-KLH IgG titers at a time point consistent with the expected timing for antibody responses following immunization. The primary time point for the analysis of the TDAR to KLH was Day 43. The data was presented for geometric mean ratio (MEDI4920/placebo) estimated from the dose response model.
Time Frame: Day 43
Population: As-treated Population.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Arm/Group | Placebo | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
Number analyzed (Participants) | 11 | 2 | 2 | 8 | 7 | 8 | 8 | 8
nanogram per milliliter (ng/mL) | NA [NA to NA] — Geometric mean ratio and 95% CI were not estimated for placebo, as the estimation was performed using the dose response model which only applies to participants who received MEDI4920. | 0.99 [0.96 to 1.01] | 0.96 [0.89 to 1.03] | 0.88 [0.72 to 1.08] | 0.68 [0.41 to 1.14] | 0.42 [0.18 to 0.97] | 0.22 [0.10 to 0.47] | 0.14 [0.06 to 0.32]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of signature of informed consent, throughout the treatment period, and the follow-up period (through Day 113 or early discontinuation visit).
Arm/Group | Placebo | MEDI4920 3 mg | MEDI4920 10 mg | MEDI4920 30 mg | MEDI4920 100 mg | MEDI4920 300 mg | MEDI4920 1000 mg | MEDI4920 3000 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/2 | 0/2 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/2 | 0/2 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 10/12 | 1/2 | 1/2 | 5/8 | 8/8 | 3/8 | 5/8 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | MEDI4920 3 mg (N=2) | MEDI4920 10 mg (N=2) | MEDI4920 30 mg (N=8) | MEDI4920 100 mg (N=8) | MEDI4920 300 mg (N=8) | MEDI4920 1000 mg (N=8) | MEDI4920 3000 mg (N=8)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | MEDI4920 3 mg (N=2) | MEDI4920 10 mg (N=2) | MEDI4920 30 mg (N=8) | MEDI4920 100 mg (N=8) | MEDI4920 300 mg (N=8) | MEDI4920 1000 mg (N=8) | MEDI4920 3000 mg (N=8)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 2 (2)
Oral herpes (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 1 (1) | 1 (2) | 3 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device failure (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.